CLINICAL TRIAL: NCT01342575
Title: Improvement of Trans-operatory X-ray Visualization During Anterior Cervical Surgery. Comparison of the Podalic Compression and Shoulder Traction Maneuvers
Brief Title: Improvement of Trans-operatory X-ray Visualization During Anterior Cervical Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: American British Cowdray Medical Center (Other)
Responsible Party: Principal Investigator, Galvan Ernesto Eduardo, MD, American British Cowdray Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ABC-11-02
Record Dates: First submitted 2011-04-20; First posted 2011-04-27 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Disk Disease
Keywords: ACDF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-operative maneuver group (Experimental)
  Interventions: Procedure: Intra-operative exposure maneuvers

INTERVENTIONS:
Procedure: Intra-operative exposure maneuvers — * Feet compression maneuver: Taking feet from the ankles, gentle pressure will be applied toward the cranium and maintained for 1 minute. X-rays and IONM will be performed
  * Arm traction maneuver: Holding two strips around the wrists and using a dynamometer adjusted to 8 kg per side, sustained traction will be maintained for 1 minute. X-rays and IONM will be performed.
  * Shoulder taping maneuver: Both shoulders will be pulled caudally with adhesive tape adjusted for a tension of 8 kg on each side. X-rays and IONM will be performed
  * Arm traction plus feet compression maneuvers: Simultaneous combination of both maneuvers as described before. X-rays and IONM will be performed
  * Shoulder taping plus feet compression maneuvers: Simultaneous combination of both maneuvers as described before. X-rays and IONM will be performed

SUMMARY:
The purpose of this study is to establish which of five different maneuvers could bring the best trans-operatory x-ray exposure during anterior cervical surgeries with the higher security

DETAILED DESCRIPTION:
Anterior cervical spine surgery (ACSS) is one of the most common spine surgery performed by neurosurgeons. One of the challenging aspects during ACSS is to achieve a correct visualization and identification of the lower levels specifically below the fifth and sixth cervical vertebras due to the difficulty of penetrating X-ray beams through the shoulders. Several methods such as taping the shoulders throughout the entire case or tying straps around the wrists and pulling them caudally temporally while shooting X-rays have been used trying to improve visualization during surgery. Both of these methods may cause problems such as brachial plexus injury, shoulder dislocations and peripheral nerve injuries.

The feet compression maneuver will be tested in terms of it's efficacy and security, as well as compared with four previous described maneuvers, using intra-operative neurophysiology monitoring (IONM).

50 consecutive patients programmed for elective ACSS that could meet inclusion criteria will be monitored with IONM using transcranial electric motor evoked potentials (tceMEPs), somatosensory evoked potentials (SSEPs) and spontaneous electromyography (EMG) after total endovenous anesthesia. On the operating table, a basal lateral x-ray picture and a first determination of IONM will be performed and used for comparison. Five maneuvers will be sequentially performed: 1) Feet compression, 2) Arm traction, 3) Arm traction plus feet compression combined, 4) Shoulder taping and 5) Shoulder taping plus feet compression.

All five maneuvers will be maintained for 1 min, time during IONM will test for changes in voltage amplitude and duration that potentially could be risky (risky is defined as a change in determinations more than 50% compared to basal determinations). Lateral x-rays will be performed during each maneuver to measure changes in segments visualization and levels exposed.

After all maneuvers are completed, we will proceed as the surgery was scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any stable biomechanically cervical pathology (like disk herniations, vertebral tumors, etc.), scheduled for ACSS

Exclusion Criteria:

* Any cervical pathology associated with segmental instability
* History of shoulder, arm, elbow or wrist pathology, including surgery or implants.
* Radiological signs of myelopathy by MRI or clinically detected
* Preoperative identified neurological deficit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-05 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Intra operative neurophysiological monitoring (IONM) alert | Participants will be followed for the duration of the surgical procedure, an expected average of 3-4 hours
  - Real time neurophysiological monitoring will be performed using evoked potentials during the whole case, specially registered during all five maneuvers. This continuous electrical surveillance let us identify any potential risk to spinal cord or nerves, founded like an IONM alert (defined as nerve irritation or a decrease in voltage and/or amplitude response). This is a single and immediate measurement obtained at surgery and it is a safety issue.

SECONDARY OUTCOMES:
Percent of segmental exposure on cervical spine lateral x-rays | Participants will be followed for the duration of surgical procedure, an expected average of 3-4 hours
  During surgery, on each of the five maneuvers, a lateral x-ray will be taken to assess the percent of visualization of the more inferior vertebra possible to see. At the surgical room, with the basal and the 5 experimental X-rays on hands, percent of exposure will be measured.
  Results will be recorded at the time of the surgery and presented showing any electrical change registered by IONM during the 5 maneuvers.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto E Galvan Hernandez, MD, MsC, Principal Investigator — American British Cowdray Medical Center, Neurological Center
Locations (1):
- American British Cowdray Medical Center, Neurological Center, Mexico City, D.F, Mexico

REFERENCES:
- [Background] Lee JY, Hilibrand AS, Lim MR, Zavatsky J, Zeiller S, Schwartz DM, Vaccaro AR, Anderson DG, Albert TJ. Characterization of neurophysiologic alerts during anterior cervical spine surgery. Spine (Phila Pa 1976). 2006 Aug 1;31(17):1916-22. doi: 10.1097/01.brs.0000228724.01795.a2. PMID 16924208
- [Background] Schwartz DM, Sestokas AK, Hilibrand AS, Vaccaro AR, Bose B, Li M, Albert TJ. Neurophysiological identification of position-induced neurologic injury during anterior cervical spine surgery. J Clin Monit Comput. 2006 Dec;20(6):437-44. doi: 10.1007/s10877-006-9032-1. Epub 2006 Sep 8. PMID 16960753
- [Background] Collado-Corona MA, de Leo-Vargas R, Sandoval-Sanchez V, Diaz-Hernandez A, Gutierrez-Sougarret BJ, Shkurovich-Bialik P. Neurophysiological monitoring in spinal cord surgery. Cir Cir. 2009 Sep-Oct;77(5):385-90. PMID 19944028